CLINICAL TRIAL: NCT03756922
Title: A Phase 1/2, Drug-Drug Interaction Study of FDL169 and FDL176 in Healthy Subjects and in Cystic Fibrosis Subjects Homozygous for the F508del-CFTR Mutation
Brief Title: A DDI Study of FDL169 and FDL176 in Healthy Subjects
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: FDL169-2018-10
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Parallel for Part 1 and Part 2; Sequential for Part 3 and Part 4
Who Masked: Participant, Care Provider, Investigator
Masking Description: Parts 1, 2, and 3 are Open Label, while Part 4 is randomized and blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): To receive a single dose of FDL176 on Day 1, followed by FDL169 TID for 28 days starting on Day 29; and another single dose of FDL176 on Day 42.
  Interventions: Drug: FDL169; Drug: FDL176
- Part 2 (Experimental): To receive FDL169 TID for 3 days from Day 1, followed by FDL176 QD for 19 days starting on Day 8; and FDL169 TID for 3 days from Day 24.
  Interventions: Drug: FDL169; Drug: FDL176
- Part 3 (Experimental): FDL169 and FDL176 for 28 days and 4 weeks of follow-up
  Interventions: Drug: FDL169; Drug: FDL176
- Part 4 (Experimental): FDL169 and FDL176 for 28 days and 4 weeks of follow-up
  Interventions: Drug: FDL169; Drug: FDL176

INTERVENTIONS:
Drug: FDL169 — CFTR corrector
Drug: FDL176 — CFTR potentiator

SUMMARY:
A DDI study to assess the safety, tolerability and pharmacokinetics of both; doses of FDL176 with and without co-administration of FDL169 and doses of FDL169 with and without co-administration of FDL176.

DETAILED DESCRIPTION:
This is an open-label, non-randomised study. Enrolment will be in two parallel and independent parts. Part 1 will assess the safety, tolerability and pharmacokinetics of single doses of FDL176 with and without co-administration of FDL169. Part 2 will assess the safety, tolerability and pharmacokinetics of repeated doses of FDL169 with and without co-administration of FDL176.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Must agree to follow the study's contraception requirement

Exclusion Criteria:

* Prior or ongoing medical condition, medical history, physical findings, ECG findings or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the subject or would place the subject at increased risk.
* History of long QT syndrome and/or QT corrected according to Fridericia's formula (QTcF) interval (>450 msec) or QTcF >450 msec at Screening or Day -1.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active.
* Use of any prescription drugs within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP.
* Use of any non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP.
* Use of any prescription and non-prescription medications that are strong inhibitors or moderate inducers of cytochrome P450 3A, within 14 days or 5-half-lives (whichever is longer) before the first dose of IMP. Use of any prescription and non-prescription medications that are strong inducers of cytochrome P450 3A within 28 days before the first dose of IMP.
* Participation in another clinical trial involving receipt of an IMP within the past 90 days.
* Prior exposure to FDL169 or FDL176
* Alkaline phosphatase, aspartate aminotransferase and/or alanine aminotransferase >1.5 x upper limit of normal (ULN) at screening.
* Serum creatinine or total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Abnormal renal function at screening, defined as estimated glomerular filtration rate <60 mL/min using the Modification of Diet in Renal Disease (MDRD) equation.
* History of human immunodeficiency virus (HIV) or positive HIV, hepatitis B or hepatitis C results at screening.
* Positive urinary drugs of abuse screen at Screening or Day -1, or positive alcohol breath test at Screening or Day -1. Consumption of alcohol within 24 h prior to admission.
* Consumption of any food or drink containing grapefruit, or Seville oranges (including marmalade and fruit juices) for 14 days before the first dose of IMP.
* Consumptions or foods containing poppy seeds or involvement in strenuous exercise for 3 days before admission.
* Known hypersensitivity to any component of the formulation of FDL169 or FDL176.
* Pregnant or nursing females.
* History of regular alcohol consumption within 6 months of the study
* Current smoking or use of tobacco products or substitutes.
* Poor peripheral venous access.
* Donation of ≥470 mL blood or loss of blood during surgery or due to trauma within 3 months prior to Day 1.
* Plasma donation within 7 days prior to Day 1.
* Failure to satisfy the Investigator of their fitness to participate for any other reason.
* Site staff, Sponsor staff or first degree family members of site or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, Cmax | Part 1: 14 weeks; Part 2: 12 weeks; Part 3: 12weeks; Part 4: 12 weeks
  Part 1: the pharmacokinetic parameters of FDL176 when co-administered with FDL169, compared to the pharmacokinetics of FDL176 alone. Part 2: the pharmacokinetics of FDL169 when co-administered with FDL176, compared to the pharmacokinetics of FDL169 alone. Part 3: PK when co-administered. Part 4: Safety and tolerability with multiple dose co-administration in CF subjects

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Part 1: 14 weeks; Part 2: 12 weeks; Part 3: 12weeks; Part 4: 12 weeks
  Safety and tolerability when FDL176 and FDL169 are co-administrated,compared to FDL176 alone, and FDL169 alone, as determined by the incidence of adverse events (Aes) and serious adverse events (SAE)s. Part 4: Combination PK and CF transmembrane conductance regulator activity in CF subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion GB Ltd, Belfast, United Kingdom